CLINICAL TRIAL: NCT00721006
Title: Phase II Safety/Efficacy Study of A Combination Stem Cell Therapy That Develops Mature Stable Vessel Formation in Ischemic Limbs
Brief Title: Phase II Combination Stem Cell Therapy for the Treatment of Severe Leg Ischemia
Acronym: MESENDO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TCA Cellular Therapy (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008-01-II
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2010-09

CONDITIONS: Critical Limb Ischemia; Severe Leg Ischemia; Peripheral Artery Disease; Peripheral Vascular Disease
Keywords: peripheral artery disease; peripheral vascular disease; PAD; PVD
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MESENDO (Experimental): All subjects will receive active treatment in a blinded fashion in the left or right lower limb. The opposite lower limb will receive placebo.
  Interventions: Biological: MESENDO
- placebo (Placebo Comparator): All subjects will receive placebo injections in a blinded fashion in the left or right lower limb. The opposite lower limb will receive active stem cell infusion
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MESENDO — 40 subcutaneous injections of biological product
  Arms: MESENDO
Biological: Placebo — 40 subcutaneous injections of placebo
  Arms: placebo

SUMMARY:
The purpose of this research study is to compare in patients with double-sided claudication if the transplant of a combination of stem cells obtained from the bone marrow of the same patient will contribute to the formation of new blood vessels in one of the severly diseased ischemic limbs(legs)versus the control limb that receives a placebo product.

Limb Ischemia (LI) is a severe obstruction of the arteries which seriously decrease blood flow to the extremities (mainly feet and legs) and has progressed to the point of severe pain and even skin ulcers or sores.

LI needs comprehensive treatment since the condition will not improve on its own. The overall goal of treatment is to reduce pain and increase blood flow to improve symptoms or save the leg and feet. In many cases, current options for treatment including medications, surgery or endovascular procedures have not been successful.

In the last few years, investigators have explored therapies aimed to increase blood flow to the ischemic vessel by transplanting cells that will promote the development of new vessels in the diseased leg.

The study hypothesis is based on the concept that the process of formation of new blood vessels is complex and requires the participation of several types of stem cells and growth factors. The lack of any of these components will produce vessels which are immature and unable to provide appropriated blood supply to the leg.

Patients eligible to participate in the this study are those suffering from double-sided claudication with poor circulation or severe leg blockages, which are not candidates for surgical procedures.

Once the mixture of stem cells is prepared and the patient's bone marrow is ready, cells will be transplanted into the calf muscle of one the the diseased legs while the other diseased leg will receive the placebo. Clinical study to evaluate and compare the efficacy of the stem cell transplant will be performed for six months post cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Males or females older than 18 years of age.
* Limb ischemia with ABI of < 0.7 in the index lower extremity in two consecutive examinations done at least 1 week apart.
* Limb ischemia with resting ischemic pain and/or claudication at 100 meters and/or non-healing ulcers.
* Claudication
* Patients not considered candidates for surgical or percutaneous revascularization, due to poor target vessels, inability to cross total occlusions, or a morbidity which precludes general anesthesia.

Exclusion Criteria:

* Inability to provide informed consent.
* Previous angiogenic therapy.
* Known sensitivity to gentamycin and/or amphotericin B.
* Use or expected use of antineoplastic drugs.
* Any illness, which might affect the patient's survival after enrollment in the protocol.
* Any illness or significant laboratory abnormality, which in the investigator's judgment will interfere with the patient's ability to comply with the protocol, compromise the patient's safety, or interfere with the interpretation of the study results.
* No evidence of acute infection
* WBC > 15000.
* WBC < 4000.
* Serum Creatinine > 3.0 mg/dL in patients who are not in hemodialysis.
* Pregnant women or women planning to become pregnant or unwilling to use appropriate birth control methods before and 2 months after cell infusion.
* Recent myocardial infarction within 3 months prior to screening.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-06; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Enhancement of vessel formation accessed by Nuclear Perfusion Scan in critical limb ischemia. | 4 months

SECONDARY OUTCOMES:
Changes in resting leg pain identified by a Visual Analog Scale and patient safety | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel P Lasala, M.D., Principal Investigator — TCA Cellular Therapy, LLC
Locations (1):
- TCA Cellular Therapy, Covington, Louisiana, United States

REFERENCES:
- [Derived] Lasala GP, Silva JA, Minguell JJ. Therapeutic angiogenesis in patients with severe limb ischemia by transplantation of a combination stem cell product. J Thorac Cardiovasc Surg. 2012 Aug;144(2):377-82. doi: 10.1016/j.jtcvs.2011.08.053. Epub 2011 Nov 12. PMID 22079876